CLINICAL TRIAL: NCT00444834
Title: A Phase II, Multi-center, Multiple-dose, Double-blind, Randomized, Crossover Study Comparing the Pharmacodynamic Effects of a Once-daily Controlled-Release Carvedilol (CRC; Egalet® Formulation) and an Immediate-Release Carvedilol (IRC) Formulation in Patients With Primary Hypertension
Brief Title: A Study of Controlled-Release Carvedilol Compared to Immediate-Release Carvedilol in Patients With Primary Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IMP supply
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-EG-006; EudraCT no.: 2006-006534-17
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Egalet carvedilol
  Interventions: Drug: Carvedilol
- 2 (Active Comparator): Coreg
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — 50 mg

SUMMARY:
The purpose of this study is to compare the efficacy of the Egalet® controlled release formulation to an immediate release Carvedilol tablet.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of mild or moderate primary hypertension
* Be able to tolerate a 2 week washout phase followed by a 2 week Placebo run- in phase
* Be minimum 18 years of age

Exclusion Criteria:

* Be intolerant to alfa- or beta-blockers
* Have secondary causes of hypertension
* Be taking more than two antihypertensive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The change from baseline to 3 weeks treatment in systolic blood pressure at the end of five minutes of sub-maximal exercise | 15w

SECONDARY OUTCOMES:
The change in Heart Rate from baseline to 3 weeks treatment measured at the end of five minutes of sub-maximal exercise | 15w
Safety | 15w

CONTACTS AND LOCATIONS:
Overall Officials: Christine Andersen, MSc Pharm, Study Director — Egalet A/S
Locations (2):
- Denmark (2):
  - Site 02, Esbjerg
  - Site 01, Frederiksberg